CLINICAL TRIAL: NCT02536066
Title: Daily Physical Activity After Meals -Long Term Effects on Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPPA99
Record Dates: First submitted 2015-05-21; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Blood Glucose; Blood Glucose Related Variables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): maintain usual physical activity patterns
- Intervention (Experimental): Addition of daily postprandial physical activity in addition to usual activity patterns
  Interventions: Behavioral: Postprandial physical activity

INTERVENTIONS:
Behavioral: Postprandial physical activity — Adding a minimum of 30 minutes of physical activity starting maximum 30 minutes after the last meal daily
  Arms: Intervention

SUMMARY:
The postprandial blood glucose concentration is an important risk factor for development of cardiovascular diseases and diabetes. Previous studies have shown that one bout of moderate or light post-meal physical activity effectively blunts the postprandial increase in blood glucose after carbohydrate intake. Pre-meal exercise does not generate such effect. Thus, the effect of exercise on postprandial glycemia depend on the timing of exercise. Even very light physical activity decreases postprandial glycemia when performed in the postprandial period. The purpose of this study was to investigate whether such activity performed each day for 12 weeks would influence blood variables related to glycemic control.

METHODS 40 subjects being ethnic Norwegians or of South Asian origin were randomized into an intervention or a control group. They were previously diagnosed as hyperglycemic, or with high risk of type 2 diabetes according to Ramachandran's risc score.

Control subjects were told to maintain their usual physical activity patterns during the study period, while the intervention subjects were instructed to undertake a minimum of 30 minutes of daily post-meal physical activity in addition to their usual activity patterns.

Venous blood samples were taken before and after the 12 week intervention period. Plasma was analyzed for HbA1c and for fasting and 2hour (OGTT) values of glucose, insulin and c-peptide. The subjects kept a physical activity diary, answered questionnaires and used accelerometers to determine the level of physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Hyperglycemia or high risk of type 2 diabetes due to Ramachandrans risk score

Exclusion Criteria:

* Use of hypoglycemic agents and conditions directly affecting blood glucose other than hyperglycemia per s.e. / diabetes type 2

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Hba1c | Pre and post intervention which lasts an average of 12 weeks
Change in Fasted glucose | Pre and post intervention which lasts an average of 12 weeks
Change in 2hour glucose | Pre and post intervention which lasts an average of 12 weeks
  Oral glucose tolerance test (OGTT)
Change in glucose during OGTT | Pre and post intervention which lasts an average of 12 weeks
  glucose measured by finger sticks every 15. minute during the 2hour oral glucose tolerance test
Change in Physical fitness measured as heart rate during an exercise test | Measured pre and post intervention which lasts an average of 12 weeks
  Heart rate measured at the end of 10 minutes ergometer cycle test an given intensity (low) to moderate intensity)
Change in Physical fitness measured as oxygen consumption during an exercise test | Measured pre and post intervention which lasts an average of 12 weeks
  measured at the end of 10 minutes ergometer cycle test an given intensity (low) by indirect calorimetry
Change in Physical fitness measured as respiratory exchange rate during an exercise test | Measured pre and post intervention which lasts an average of 12 weeks
  Measured at the end of 10 minutes ergometer cycle test an given intensity (low), by indirect calorimetry
Change in Physical fitness measured as perceived exertion during an exercise test | Measured pre and post intervention which lasts an average of 12 weeks
  Borg RPE scale measured at the end of 10 minutes ergometer cycle test an given intensity (low)
Change in Physical fitness measured as lactic acid during an exercise test | Measured pre and post intervention which lasts an average of 12 weeks
  measured at the end of 10 minutes ergometer cycle test an given intensity (low) from capillary blod from a finger stick

SECONDARY OUTCOMES:
Change in Total cholesterol | Measured Pre and post intervention which lasts an average of 12 weeks
Change in LDL cholesterol | Measured Pre and post intervention which lasts an average of 12 weeks
Change in HDL cholesterol | Measured Pre and post intervention which lasts an average of 12 weeks
Change in triglycerides | Measured Pre and post intervention which lasts an average of 12 weeks
Change in body weight | Measured Pre and post intervention which lasts an average of 12 weeks
Change in waist circumference | Measured Pre and post intervention which lasts an average of 12 weeks
Change in Blood pressure | Measured Pre and post intervention which lasts an average of 12 weeks
Change in Quality of life | Measured Pre and post intervention which lasts an average of 12 weeks
  Quality of life measured by SF36

OTHER OUTCOMES:
Change in Level of physical activity | Measured for 4 days pre intervention and 4 days in the middle of intervention
  Measured by accelerometer
Change in dietary habits | Measured for 4 days pre intervention and 4 days in the middle of intervention
  Measured by dietary registration with dietary diary and a kitchen scale

CONTACTS AND LOCATIONS:
Overall Officials: håvard nygaard, msc, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Lillehammer University College, Lillehammer, Norway